CLINICAL TRIAL: NCT02549339
Title: Efficacy and Safety of LEO 43204 in the Field Treatment of Actinic Keratosis on Face or Chest Including 12-month Follow-up
Brief Title: Efficacy and Safety of LEO 43204 in the Field Treatment of Actinic Keratosis on Face or Chest including12-month Follow-up
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LP0084-1194
Record Dates: First submitted 2015-09-09; First posted 2015-09-15 (Estimated); Results first posted 2018-11-14 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2018-10

CONDITIONS: Actinic Keratosis
MeSH Terms: conditions — Keratosis, Actinic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- LEO 43204 gel (Experimental): Treatment once daily for 3 days
  Interventions: Drug: LEO 43204 gel
- Vehicle gel (Placebo Comparator): Treatment once daily for 3 days
  Interventions: Drug: Vehicle gel

INTERVENTIONS:
Drug: LEO 43204 gel
  Arms: LEO 43204 gel
Drug: Vehicle gel
  Arms: Vehicle gel

SUMMARY:
The objective of the trial is to compare the short term efficacy of LEO 43204 gel with vehicle gel in AK on face or chest when applied topically once daily for 3 consecutive days as field treatment

ELIGIBILITY:
Inclusion Criteria:

* Subjects with 5 to 20 clinically typical, visible and discrete AKs within a treatment area of sun-damaged skin on either the full face or a contiguous area of approximately 250 cm2 (40 in2) on the chest
* Subjects with minimum 3 clinically typical, visible and discrete AKs within a tracking area of 50 cm2 (8 in2). The tracking area must be within the treatment area

Exclusion Criteria:

* Location of the treatment area (full face or chest) within 5 cm of an incompletely healed wound or within 5 cm of a suspected BCC or SCC
* Treatment with ingenol mebutate gel in the treatment area within the last 12 months
* Lesions in the treatment area that have: atypical clinical appearance (e.g. hyperthrophic, hyperkeratotic or cutaneous horns) and /or, recalcitrant disease (e.g. did not respond to cryotherapy on two previous occasions)
* History or evidence of skin conditions other than the trial indication that would interfere with the evaluation of the trial medication (e.g., eczema, unstable psoriasis, xeroderma pigmentosum)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 383 (Actual)
Dates: Start 2015-11-13 (Actual); Primary Completion 2016-08-05 (Actual); Study Completion 2017-08-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: C. William Hanke, MD, Principal Investigator — Laser & Skin Surgery Center of Indiana
Locations (1):
- Laser & Skin Surgery Center of Indiana, Carmel, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Clinical Trials at LEO Pharma — https://www.leopharmatrials.com/en

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 383 participants were enrolled across 5 countries: United States, Canada, Germany, Spain, and Italy. 74 were screening failures, and 309 participants were randomized to 1 of the 2 treatment groups.
Groups:
- LEO 43204 0.018% Gel: Treatment with LEO 43204 0.018% gel once daily for 3 consecutive days applied on full face or within a contiguous area of approximately 250 cm2 on the chest.
- Vehicle Gel: Treatment with vehicle gel once daily for 3 consecutive days applied on full face or within a contiguous area of approximately 250 cm2 on the chest.
Period: 3-day Treatment and 8-week Follow-up
Arm/Group | LEO 43204 0.018% Gel | Vehicle Gel
Started | 205 | 104
Treated | 202 | 104
Completed | 201 | 99
Not Completed | 4 | 5
Not completed — Protocol Violation | 2 | 0
Not completed — Withdrawal by Subject | 1 | 3
Not completed — Other | 1 | 0
Not completed — Lost to Follow-up | 0 | 2
Period: 12-month Follow-up
Arm/Group | LEO 43204 0.018% Gel | Vehicle Gel
Started | 201 | 98
Completed | 192 | 87
Not Completed | 9 | 11
Not completed — Lack of Efficacy | 0 | 2
Not completed — Withdrawal by Subject | 8 | 3
Not completed — Lost to Follow-up | 1 | 3
Not completed — Other | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- LEO 43204 0.018% Gel: Treatment once daily for 3 days with LEO 43204 0.018% gel
- Vehicle Gel: Treatment once daily for 3 days with vehicle gel
- Total: Total of all reporting groups
Arm/Group | LEO 43204 0.018% Gel | Vehicle Gel | Total
Number analyzed (Participants) | 202 | 104 | 306
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.1 (9.2) | 66.3 (9.1) | 68.2 (9.3)
Age, Customized [Count of Participants; unit: Participants]
  Age group: 18-64 years | 63 | 38 | 101
  Age group: 65-84 years | 131 | 65 | 196
  Age group: >=85 years | 8 | 1 | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65 | 41 | 106
  Male | 137 | 63 | 200
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 103 | 55 | 158
  Canada | 47 | 26 | 73
  Germany | 26 | 10 | 36
  Spain | 14 | 7 | 21
  Italy | 12 | 6 | 18

OUTCOME MEASURES:

1. Primary Outcome: Complete Clearance of Actinic Keratosis (AK)
Description: The number of clinically visible actinic keratosis lesions (AKs) identified in the treatment area was recorded at Day 1, Week 4, and Week 8.
  Complete clearance was defined as no clinically visible AKs in the treatment area.
  The table shows the percentage of mean number of subjects across imputations with complete clearance.
Time Frame: At Week 8
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | LEO 43204 0.018% Gel | Vehicle Gel
Number analyzed (Participants) | 202 | 104
percentage of participants | 20.4 [14.9 to 26.0] | 2.9 [-0.3 to 6.1]
Statistical Analysis 1: Comparison: LEO 43204 0.018% Gel vs Vehicle Gel; Test type: Superiority; p = 0.001, Mantel Haenszel; Ratio of clearance rates = 7.57, 95% CI 2-sided [2.26 to 25.31] — Mantel-Haenszel estimate (0.018% relative to vehicle), adjusted for pooled sites

2. Secondary Outcome: Percentage of Participants With Partial Clearance (Multiple Imputation)
Description: The number of clinically visible AKs identified in the treatment area was recorded at Day 1, Week 4, and Week 8.
  Partial clearance was defined as at least 75% reduction from baseline in the number of clinically visible AKs in the treatment area.
  The table shows the percentage of mean number of participants across imputations with partial clearance.
Time Frame: At Week 8
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | LEO 43204 0.018% Gel | Vehicle Gel
Number analyzed (Participants) | 202 | 104
percentage of participants | 60.3 [53.5 to 67.1] | 10.7 [4.7 to 16.7]
Statistical Analysis 1: Comparison: LEO 43204 0.018% Gel vs Vehicle Gel; The p-values for secondary endpoints have been corrected by the Holm-Bonferroni method to account for multiplicity. The prespecified multiplicity adjustment by the Holm-Bonferroni method requires the ordering of the p-values for the secondary endpoints by size; Test type: Superiority; p < 0.001, Mantel Haenszel; Ratio of clearance rates = 5.90, 95% CI 2-sided [3.30 to 10.54] — Mantel-Haenszel estimate (0.018% relative to vehicle), adjusted for pooled sites

3. Secondary Outcome: Percentage of Participants With Partial Clearance (Multiple Imputation)
Description: as for outcome 2
Time Frame: At Week 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | LEO 43204 0.018% Gel | Vehicle Gel
Number analyzed (Participants) | 202 | 104
percentage of participants | 61.1 [54.4 to 67.8] | 10.8 [4.8 to 16.9]
Statistical Analysis 1: Comparison: LEO 43204 0.018% Gel vs Vehicle Gel; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p < 0.001, Mantel Haenszel; Ratio of clearance rates = 5.75, 95% CI 2-sided [3.24 to 10.20] — Mantel-Haenszel estimate (0.018% relative to vehicle), adjusted for pooled sites

4. Secondary Outcome: Percent Reduction in AK Count in the Treatment Area Compared to Baseline
Description: The percent reduction at Week 8 from baseline was analysed using a negative binomial regression for the AK count at Week 8 with treatment group and pooled sites as factors and baseline count as offset variable (using multiple imputations to account for missing values). The table presents adjusted mean percent reduction at Week 8 from baseline.
Time Frame: At Week 8
Measure: Mean (95% Confidence Interval); unit: percentage of reduction
Arm/Group | LEO 43204 0.018% Gel | Vehicle Gel
Number analyzed (Participants) | 202 | 104
percentage of reduction | 74.8 [71.8 to 77.4] | 15.0 [3.4 to 25.2]
Statistical Analysis 1: Comparison: LEO 43204 0.018% Gel vs Vehicle Gel; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p < 0.001, Mantel Haenszel — Negative binominal regression with treatment group and pooled site as factors and log baseline count as offset variable; Week 8 AK count ratio = 0.30, 95% CI 2-sided [0.25 to 0.35] — 0.018% relative to vehicle

ADVERSE EVENTS:
Time Frame: Treatment period including follow-up (from Day 1 to Week 8) and extended follow-up (from Week 8 up to Month 14)
Description: Adverse events presented in the table are investigator-reported terms.
  Adverse events of special interest within system organ class (SOC) Neoplasm benign, malignant and unspecified (incl cysts and polyps), were adjudicated by an Independent Adjudication Committee based on central biopsy review.
  For further details on the adjudication outcomes, see link to the full report in section "More information"
Groups:
- LEO 43204 0.018% Gel; LEO 43204 0.018% Gel - Extended Follow-up: Treatment once daily for 3 days LEO 43204 0.018% gel
- Vehicle Gel; Vehicle Gel - Extended Follow-up: Treatment once daily for 3 days Vehicle gel
Arm/Group | LEO 43204 0.018% Gel | Vehicle Gel | LEO 43204 0.018% Gel - Extended Follow-up | Vehicle Gel - Extended Follow-up
Serious Adverse Events (participants affected / at risk) | 0/202 | 0/104 | 1/201 | 0/98
Other Adverse Events (participants affected / at risk) | 136/202 | 32/104 | 35/201 | 14/98
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LEO 43204 0.018% Gel (N=202) | Vehicle Gel (N=104) | LEO 43204 0.018% Gel - Extended Follow-up (N=201) | Vehicle Gel - Extended Follow-up (N=98)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 — The event was classified as serious because the participant was hospitalized.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LEO 43204 0.018% Gel (N=202) | Vehicle Gel (N=104) | LEO 43204 0.018% Gel - Extended Follow-up (N=201) | Vehicle Gel - Extended Follow-up (N=98)
Application site pain (General disorders) | 113 | 5 | 0 | 0
Application site pruritus (General disorders) | 63 | 5 | 0 | 1
Application site discomfort (General disorders) | 9 | 3 | 0 | 0
Application site warmth (General disorders) | 3 | 1 | 0 | 0
Application site paraesthesia (General disorders) | 2 | 1 | 0 | 0
Chills (General disorders) | 3 | 0 | 0 | 0
Pain (General disorders) | 1 | 1 | 0 | 0
Application site dryness (General disorders) | 1 | 0 | 0 | 0
Application site haematoma (General disorders) | 0 | 1 | 0 | 0
Application site laceration (General disorders) | 0 | 1 | 0 | 0
Application site nodule (General disorders) | 1 | 0 | 0 | 0
Chest discomfort (General disorders) | 1 | 0 | 0 | 0
Facial pain (General disorders) | 1 | 0 | 0 | 0
Hangover (General disorders) | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 0 | 0
Periorbital oedema (Eye disorders) | 8 | 0 | 0 | 0
Eye irritation (Eye disorders) | 4 | 1 | 0 | 0
Lacrimation increased (Eye disorders) | 2 | 1 | 0 | 0
Eye pain (Eye disorders) | 2 | 0 | 0 | 0
Conjunctival haemorrhage (Eye disorders) | 0 | 1 | 0 | 0
Dry eye (Eye disorders) | 1 | 0 | 0 | 0
Eczema eyelids (Eye disorders) | 1 | 0 | 0 | 0
Eyelid oedema (Eye disorders) | 1 | 0 | 0 | 0
Eyelid pain (Eye disorders) | 1 | 0 | 0 | 0
Photophobia (Eye disorders) | 1 | 0 | 0 | 0
Vision blurred (Eye disorders) | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 6 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 3 | 1 | 0 | 0
Rhinitis (Infections and infestations) | 3 | 0 | 0 | 0
Herpes simplex (Infections and infestations) | 2 | 0 | 1 | 1
Application site infection (Infections and infestations) | 1 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 1 | 0 | 0 | 0
Folliculitis (Infections and infestations) | 0 | 1 | 0 | 0
Furuncle (Infections and infestations) | 0 | 1 | 0 | 0
Influenza (Infections and infestations) | 1 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 4 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0
Accidental exposure to product (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Face injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Periorbital haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Sunburn (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 3 | 9 | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 0 | 6 | 3
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 10 | 2
Headache (Nervous system disorders) | 12 | 0 | 0 | 0
Anosmia (Nervous system disorders) | 1 | 0 | 0 | 0
Sciatica (Nervous system disorders) | 1 | 0 | 0 | 0
Tension headache (Nervous system disorders) | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
Exostosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Rectal polyp (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 3 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0 | 0
Sleep disorder (Psychiatric disorders) | 1 | 0 | 0 | 0
Prostatitis (Reproductive system and breast disorders) | 2 | 0 | 0 | 0
Prostatomegaly (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Intertrigo (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Post inflammatory pigmentation change (Skin and subcutaneous tissue disorders) | 0 | 1 | 4 | 1
Blood creatinine increased (Investigations) | 1 | 0 | 0 | 0
Liver function test abnormal (Investigations) | 1 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0 | 0
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 2
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 3 | 0
Hypertrophic scar (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0
Papule (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Rosacea (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Application site scar (General disorders) | 0 | 0 | 3 | 3
Application site discolouration (General disorders) | 0 | 0 | 1 | 1
Application site dermatitis (General disorders) | 0 | 0 | 1 | 0
Application site macule (General disorders) | 0 | 0 | 0 | 1
Postoperative wound infection (Infections and infestations) | 0 | 0 | 1 | 0
Scar (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
LEO acknowledges the investigators right to publish the entire results of the study, irrespective of outcome. LEO retains the right to have any publication submitted to LEO for review. Investigators must undertake not to submit any part of their individual data for publication without the prior consent of LEO.